CLINICAL TRIAL: NCT04156841
Title: Sentinel Lymph Node Biopsy in Early Breast Cancer: a Real-world Multicenter Cross-sectional Study (CABS001 Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20192114-C-1
Record Dates: First submitted 2019-09-29; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- performed SLNB using a single mapping agent
  Interventions: Diagnostic Test: mapping agent
- performed SLNB by combination of blue dye and radiotracer
  Interventions: Diagnostic Test: mapping agent
- underwent SLN surgery receiving neoadjuvant chemotherapy
  Interventions: Procedure: neoadjuvant chemotherapy
- underwent SLN surgery not receiving neoadjuvant chemotherapy
  Interventions: Procedure: neoadjuvant chemotherapy

INTERVENTIONS:
Diagnostic Test: mapping agent — according to different tracer methods, patients are divided into the implementation of a single mapping agent and implementation of combination of blue dye and radiotracer agent.
  Groups: performed SLNB by combination of blue dye and radiotracer; performed SLNB using a single mapping agent
Procedure: neoadjuvant chemotherapy — Patients were divided into two groups based on whether they were receiving neoadjuvant chemotherapy.
  Groups: underwent SLN surgery not receiving neoadjuvant chemotherapy; underwent SLN surgery receiving neoadjuvant chemotherapy

SUMMARY:
Objective: To investigate the current clinical practice of sentinel lymph node biopsy (SLNB) in patients with early stage breast cancer in China. Methods: The data of early breast cancer patients who underwent SLNB in 40 Grade III Level A hospitals in China in 2018 will be collected. Different centers, tracer methods, molecular typing and neoadjuvant chemotherapy will be used as stratification factors to analyze the implementation rate, number of detections, positive rate of SLNB and the follow-up treatment.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer confirmed by fine needle aspiration or biopsy
* SLNB with or without axillary lymph node dissection
* receiving conventional systematic treatment or regional treatment
* complete medical record.

Exclusion Criteria:

* IV stage breast cancer
* combined with secondary invasive malignant tumor
* diagnosed with other serious disease, including congestive heart failure (NYHA cardiac function grade II, III, IV) or congestive heart failure, unstable angina pectoris, myocardial infarction, high-risk uncontrollable heart rate disorder or other serious cardiovascular diseases within 6 months
* difficulty breathing at rest or need oxygen therapy
* severe infection
* uncontrolled diabetes
* serious psychological or mental disorders
* poor compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: early breast cancer patients who underwent SLNB in 40 Grade III Level A hospitals in China in 2018
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the performance rate of sentinel lymph node biopsy (SLNB) in patients with early stage breast cancer in China | 2020-12-31
  the performance rate of SLNB refers to the number of patients implementing SLNB divided by the total number of breast cancer patients
the positive rate of SLNs in patients with early stage breast cancer in China | 2020-12-31
  SLNs positive rate is the number of positive SLN patients divided by the number of patients implementing SLNB
the number of resected SLNs in patients with early stage breast cancer in China | 2020-12-31
  the average number of resected SLNB will be calculated

SECONDARY OUTCOMES:
incidence of infection events after SLNB in patients with early stage breast cancer in China | 2021-12-31
  incidence of infection events is the number of patients who have an infection event after SLNB divided by the total number of patients implementing SLNB. The infection events include incision infection, local skin infection and injured vascular infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No